CLINICAL TRIAL: NCT00432978
Title: Effect of Bosentan on Exercise Capacity at High Altitude
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VA Loma Linda Health Care System (U.S. Federal Agency)
Collaborators: Actelion (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 00534; Prom: 0030
Record Dates: First submitted 2007-02-06; First posted 2007-02-08 (Estimated); Last update posted 2007-04-18 (Estimated); Status verified 2007-04

CONDITIONS: Altitude; Pulmonary Hypertension
Keywords: hypoxia; endothelin; exercise
MeSH Terms: conditions — Hypertension, Pulmonary; Hypoxia; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Bosentan administration

SUMMARY:
This study is to determine whether bosentan will alter exercise capacity after rapid ascent to high altitude.

We hypothesize that bosentan administration will improve arterial oxygenation and exercise capacity.

DETAILED DESCRIPTION:
Both the prostacyclin and the nitric oxide pathways are important in modulating hypoxic pulmonary vasoconstriction (HPV). There is little information about the role of the endothelin pathway at high altitude. The endothelin pathway involves the activation of two distinct receptors, A and B. Bosentan is a nonpeptide, specific, competitive, dual antagonist of both endothelin receptor subtypes. The primary objective of this study will be to determine the effect of endothelin receptor blockade with bosentan on exercise performance and HPV. This is a prospective, double blind, placebo-controlled, randomized cross-over study involving healthy subjects aged 25-55 years of age. Subjects will undergo echocardiography and exercise testing at low altitude (< 500m) and at 3800m. Subjects will receive either bosentan vs. placebo and will be studied at low and high altitude on two occasions in a crossover design. Primary outcome measures will be pulmonary artery systolic pressure measured by echo-Doppler and exercise capacity. A better understanding of the role of the endothelin pathway in HPV may lead to improved treatments for some patients.

ELIGIBILITY:
Inclusion Criteria:

* Normal healthy subjects aged 18 - 55 years

Exclusion Criteria:

* Pregnancy
* Heart, lung or liver disease
* Use of glyburide, cyclosporin A

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20
Dates: Start 2006-07; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Exercise Capacity
Pulmonary artery systolic pressure

SECONDARY OUTCOMES:
Hemoglobin oxygen saturation

CONTACTS AND LOCATIONS:
Overall Officials: James D Anholm, MD, Principal Investigator — VA Loma Linda Healthcare System; Katja Ruh, MD, Principal Investigator — Loma Linda University
Locations (1):
- VA Loma Linda Healthcare System, Loma Linda, California, United States

REFERENCES:
- [Derived] Seheult RD, Ruh K, Foster GP, Anholm JD. Prophylactic bosentan does not improve exercise capacity or lower pulmonary artery systolic pressure at high altitude. Respir Physiol Neurobiol. 2009 Feb 28;165(2-3):123-30. doi: 10.1016/j.resp.2008.10.005. Epub 2008 Oct 11. PMID 18977464